CLINICAL TRIAL: NCT02353884
Title: Multi-modality MRI Study on Prediction for Mild Cognitive Impairment Conversion
Status: Completed | Type: Observational
Sponsor: XuanwuH 2 (Other)
Collaborators: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Chief physician, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Other Study IDs: hanying3
Record Dates: First submitted 2014-10-04; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- MCIp,MCIs: progressive MCI：those convert to AD in two years, stable MCI
- MCI，HC: mild cognitive impairment, healthy control

SUMMARY:
The purpose of this study is to find the characteristics of mild cognitive impairment (MCI) using technology of Multi-Modality MRI , including structural MRI, functional MRI and diffusion tensor imaging(DTI). Then analyze the difference between progressive MCI (MCIp) and stable MCI (MCIs) and further construct the predictable classifier from MCI to Alzheimer's disease (AD) based on Multi-Modality MRI characteristics of MCI patients.

DETAILED DESCRIPTION:
The cognition of MCI is between normal healthy and AD, which is thought the transitional stage of AD. Patients with MCI have heavy risk to convert to AD, so in this study, the investigators focus on the exploration of the characteristics of mild cognitive impairment (MCI) using technology of Multi-Modality MRI, including structural MRI, functional MRI and DTI. Then the investigators further study the patients who convert to AD and explore their MRI characteristics on baseline, in order to construct the predictable classifier from MCI to AD. The investigators want to achieve the early diagnosis of AD and help clinicians interfere with the progress of this disease.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 55 to 75 years old
* Memory loss complaint and confirmed by an informant
* Cognitive impairment in single or multiple domains, adjusted for age and education
* Normal or near-normal performance on general cognitive function and no or minimum impairment of daily life activities
* A Clinical Dementia Rating (CDR) score is 0.5 and consistent with the boundary of neuropsychological scale
* Failure to meet the criteria for dementia
* Must be able to accept examination of MRI, sight and hearing allow to complete test
* Right handedness

Exclusion Criteria:

* Other diseases that cause cognitive impairment, such as thyroid disease, stroke and so on
* People who have severe visual and hearing impairment

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cognition of MCI is between healthy control and AD, which is thought the transitional stage of AD. Patients with MCI have heavy risk to convert to AD.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
the accuracy of a predictable classifier from MCI to AD based on Multi-Modality MRI characteristics of MCI patients. | 2 years
  one-hundred MCI subjects and 50 healthy controls recruited underwent structure,resting-state functional magnetic resonance imaging and diffusion tensor imaging.After 2-year follow-up,the MCI subjects were divided into progressive MCI(MCIp) and stable MCI(MCIs).Based on differences among MCIp，MCIs and healthy controls in baseline neuroimaging data，some suitable indicators were selected，and then a predictable classifier from MCI to AD based on multi-modality MRI was constructed.At last，the leave-one-out cross validation analysis were conducted to estimate the accuracy of the classifier.The classification accuracy was measured by the proportion of MCI subjects that were correctly classified into the MCIp or MCIs groups

SECONDARY OUTCOMES:
characteristic changes of brain structure in progressive MCI | 2 years
  voxel based morphometry (VBM) and cortical-thicknessanalysis（CTA）based on structural MRI were used to characterize the changes of brain structure in the MCIp comparing with the MCIs and healthy control
characteristic changes of anatomical connectivity in progressing MCI | 2 years
  region of interest(ROI),voxel and fiber bundle analysis based on diffusion tensor imaging were used to detect differences among the MCIp，MCIs and healthy control in fractional anisotropy(FA) and mean diffusivity(MD).
characteristic changes of functional connectivity in progressing MCI | 2 years
  functional connectivity（FC） was compared among the MCIp, MCIs and healthy control using resting-state functional magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurolgy,Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Sheng C, Sun Y, Wang M, Wang X, Liu Y, Pang D, Liu J, Bi X, Du W, Zhao M, Li Y, Li X, Jiang J, Han Y. Combining Visual Rating Scales for Medial Temporal Lobe Atrophy and Posterior Atrophy to Identify Amnestic Mild Cognitive Impairment from Cognitively Normal Older Adults: Evidence Based on Two Cohorts. J Alzheimers Dis. 2020;77(1):323-337. doi: 10.3233/JAD-200016. PMID 32716355
- [Derived] Yang L, Yan Y, Wang Y, Hu X, Lu J, Chan P, Yan T, Han Y. Gradual Disturbances of the Amplitude of Low-Frequency Fluctuations (ALFF) and Fractional ALFF in Alzheimer Spectrum. Front Neurosci. 2018 Dec 20;12:975. doi: 10.3389/fnins.2018.00975. eCollection 2018. PMID 30618593